CLINICAL TRIAL: NCT03426566
Title: Prevention of Foot Injuries - Abnormal Distribution Patterns of Plantar Pressure in Patients With Diabetes and Its Connection to Peripheral Neuropathy, Gender, Age and BMI
Brief Title: Abnormal Plantar Pressure in Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Edyta Sutkowska, MD, PhD; Head of the Department and Division of Medical Rehabilitation, Wroclaw Medical University
Other Study IDs: ST 690
Record Dates: First submitted 2018-01-23; First posted 2018-02-08 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Complications
Keywords: diabetic foot; pedobarography; diabetic neuropathy; plantar pressure
MeSH Terms: conditions — Diabetes Complications; Diabetic Foot; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with diabetes: Data from medical records from : non-ulcer patients with DM (diabetes mellitus) from the Diabetic Foot Centre (DFC) in Wroclaw. As it is a retrospective analysis no intervention is planned.
  Interventions: Other: retrospective observational study with no intervention

INTERVENTIONS:
Other: retrospective observational study with no intervention — no intervention

SUMMARY:
The prevalence of abnormal plantar pressure distribution (APD) and its connection with various factors among patients with diabetes is not known. The purpose of this study was to evaluate the prevalence of the APD and its connection with selected factors among patients with diabetes.

DETAILED DESCRIPTION:
The abnormal plantar pressure distribution (APD) plays a key role in the formation of plantar calluses which are responsible for diabetic foot ulcer.

The knowledge of APD is necessary to plan proper prevention in the group of patients with diabetes mellitus (DM).

Medical records from previous patients' visits of non-ulcer patients with diabetes were retrospectively analysed. The relationship between APD, obtained during a pedobarographic test as a semi-quantitative assessment with colourful print analysis, and neuropathy, gender, age and BMI was searched.

ELIGIBILITY:
Inclusion Criteria:

* subjects with diabetes mellitus diagnosis
* citizens
* no previous foot ulceration and/or foot surgery

Exclusion Criteria:

* previous foot ulceration and/or foot surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wroclaw (where the Diabetic Foot Centre exists) citizens who came spontaneously to be examined despite the absence of diabetic foot signs or symptoms
Sampling Method: Probability Sample
Enrollment: 974 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edyta Sutkowska, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Department and Division of Medical Rehabilitation, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
all collected individual participant data but without individual foot-print picture (mostly paper documentation) ; only the example of foot -print with explanation is available
Supporting Information: Study Protocol, SAP
Time Frame: no limit
Access Criteria: will be included in an article and/or as supplementary materials

REFERENCES:
- [Background] Boulton AJ, Hardisty CA, Betts RP, Franks CI, Worth RC, Ward JD, Duckworth T. Dynamic foot pressure and other studies as diagnostic and management aids in diabetic neuropathy. Diabetes Care. 1983 Jan-Feb;6(1):26-33. doi: 10.2337/diacare.6.1.26. PMID 6839919
- [Background] Boulton AJ, Betts RP, Franks CI, Newrick PG, Ward JD, Duckworth T. Abnormalities of foot pressure in early diabetic neuropathy. Diabet Med. 1987 May-Jun;4(3):225-8. doi: 10.1111/j.1464-5491.1987.tb00867.x. PMID 2956023
- [Background] Duckworth T, Boulton AJ, Betts RP, Franks CI, Ward JD. Plantar pressure measurements and the prevention of ulceration in the diabetic foot. J Bone Joint Surg Br. 1985 Jan;67(1):79-85. doi: 10.1302/0301-620X.67B1.3968150.
- [Background] Rich J, Veves A. Forefoot and rearfoot plantar pressures in diabetic patients: correlation to foot ulceration. Wounds2000;12:82-87
- [Background] Frykberg RG, Lavery LA, Pham H, Harvey C, Harkless L, Veves A. Role of neuropathy and high foot pressures in diabetic foot ulceration. Diabetes Care. 1998 Oct;21(10):1714-9. doi: 10.2337/diacare.21.10.1714. PMID 9773736
- [Background] Bakker K, Schaper NC; International Working Group on Diabetic Foot Editorial Board. The development of global consensus guidelines on the management and prevention of the diabetic foot 2011. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:116-8. doi: 10.1002/dmrr.2254. PMID 22271736
- [Background] Choi YR, Lee HS, Kim DE, Lee DH, Kim JM, Ahn JY. The diagnostic value of pedobarography. Orthopedics. 2014 Dec;37(12):e1063-7. doi: 10.3928/01477447-20141124-52. PMID 25437079
- [Background] Bakker K, Apelqvist J, Lipsky BA, Van Netten JJ; International Working Group on the Diabetic Foot. The 2015 IWGDF guidance documents on prevention and management of foot problems in diabetes: development of an evidence-based global consensus. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:2-6. doi: 10.1002/dmrr.2694. PMID 26409930
- [Background] Crawford F, Cezard G, Chappell FM, Murray GD, Price JF, Sheikh A, Simpson CR, Stansby GP, Young MJ. A systematic review and individual patient data meta-analysis of prognostic factors for foot ulceration in people with diabetes: the international research collaboration for the prediction of diabetic foot ulcerations (PODUS). Health Technol Assess. 2015 Jul;19(57):1-210. doi: 10.3310/hta19570. PMID 26211920
- [Background] Inlow S. The 60-second Foot Exam for People with Diabetes. Wound Care Can2004;2:10-11
- [Background] Carreau L, Niezgoda H, LeBlond S, Trainor A, Orsted H, Woodbury MG. A prospective, descriptive study to assess the reliability and usability of a rapid foot screen for patients with diabetes mellitus in a complex continuing care setting. Ostomy Wound Manage. 2013 Jan;59(1):28-34. PMID 23308404
- [Background] Tuna H, Birtane M, Güldiken S et al. The effect of disease duration on foot plantar pressure values in patients with type 2 diabetes mellitus. Turk J Phys Med Rehab2014;60:231-235
- [Background] Lazaro-Martinez JL, Aragon-Sanchez FJ, Beneit-Montesinos JV, Gonzalez-Jurado MA, Garcia Morales E, Martinez Hernandez D. Foot biomechanics in patients with diabetes mellitus: doubts regarding the relationship between neuropathy, foot motion, and deformities. J Am Podiatr Med Assoc. 2011 May-Jun;101(3):208-14. doi: 10.7547/1010208. PMID 21622632
- [Background] Perell KL, Merrill V, Nouvong A. Location of plantar ulcerations in diabetic patients referred to a Department of Veterans Affairs podiatry clinic. J Rehabil Res Dev. 2006 Jul-Aug;43(4):421-6. doi: 10.1682/jrrd.2005.10.0157. PMID 17123181
- [Background] Ledoux WR, Shofer JB, Cowley MS, Ahroni JH, Cohen V, Boyko EJ. Diabetic foot ulcer incidence in relation to plantar pressure magnitude and measurement location. J Diabetes Complications. 2013 Nov-Dec;27(6):621-6. doi: 10.1016/j.jdiacomp.2013.07.004. Epub 2013 Sep 4. PMID 24012295
- [Background] Hills AP, Hennig EM, McDonald M, Bar-Or O. Plantar pressure differences between obese and non-obese adults: a biomechanical analysis. Int J Obes Relat Metab Disord. 2001 Nov;25(11):1674-9. doi: 10.1038/sj.ijo.0801785. PMID 11753590
- [Background] Sutkowska E, Fortuna P, Kaluza B, Sutkowska K, Hodurek P, Fleszar MG. The impact of Sample Handling Time on metformin serum concentration. Biomed Pharmacother. 2021 Jan;133:110971. doi: 10.1016/j.biopha.2020.110971. Epub 2020 Nov 25. PMID 33248407
- [Result] Sutkowska E, Sutkowski K, Sokolowski M, Franek E, Dragan S Sr. Distribution of the Highest Plantar Pressure Regions in Patients with Diabetes and Its Association with Peripheral Neuropathy, Gender, Age, and BMI: One Centre Study. J Diabetes Res. 2019 Jul 9;2019:7395769. doi: 10.1155/2019/7395769. eCollection 2019. PMID 31380446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: between October 2009 and December 2010 Medical records were obtained from the Diabetic Foot Centre (DFC) in Wroclaw, Poland and covered a period of fifteen months of work.
Pre-assignment Details: Patients without previous ulcerations or foot surgery were evaluated.
Units Other Than Participants: feet
Period: Overall Study
Arm/Group | Patients With Diabetes
Started | 974; 1948 feet
Completed | 974; 1948 feet
Not Completed | 0; 0 feet

BASELINE CHARACTERISTICS:
Units Other Than Participants: feet
Arm/Group | Patients With Diabetes
Number analyzed (Participants) | 974
Number analyzed (feet) | 1948
Age, Categorical [Count of Participants; unit: Participants] — Age- was calculated based on patients identification (ID) number (in Poland each ID number contains date of birth).
  Participants
    <=18 years | 0
    Between 18 and 65 years | 478
    >=65 years | 496
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 523
  Male | 451
Region of Enrollment [Number; unit: participants]
  Poland | 974

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Plantar Pressure Distribution
Description: static pedobarographic test with semi-quantitative assessment: number of the patients with abnormal plantar pressure location based on a semi-quantitative method, as static barefoot pedobarographic records with colourful print analysis. The intensity of colour was proportional to the pressure received. Warm colours indicated the greatest pressure, while cold colours indicated the least plantar pressure (starting with red, then yellow, green, and blue)
Time Frame: 1 visit
Population: Patients with diabetes mellitus but without active or past foot ulcer or surgical procedure within the feet. Abnormal plantar pressure distribution (APD) - means number of participants with symmetrical abnormal pressure distribution; No APD- without such kind a distribution.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Diabetes: Patients with diabetes from Diabetic Foot Centre
Arm/Group | Patients With Diabetes
Number analyzed (Participants) | 974
Participants
  patients without APD | 80
  patients with APD | 894

2. Secondary Outcome: Number of Participants With Positive Test for Neuropathy
Description: Peripheral neuropathy is assessed with questions and clinical evaluation. A nurse asks the patient about stinging, numbness, tingling, or burning of the foot. Ten-gram monofilament and tuning fork (128 MHz) tests are administered. Monofilament is applied in 10 locations on the sole and one on the dorsal part of the foot for checking the loss of protective sensation. A positive monofilament test is considered to be the lack of sensation of tightness in at least 6 of 11 tested sites. The tuning fork is applied for vibration detection to both ankles, the first metatarsophalangeal joint, and the anterior aspect of the shin bone sites. A positive vibration test is considered to be no detection of vibration in three of four test sites.Two positive test results and typical symptoms of neuropathy are the basis for confirmation of peripheral symmetric sensory neuropathy (PSSN). The condition required for the occurrence of these disorders was symmetry.
Time Frame: 1 visit
Population: Patients with DM, without active or past ulcer or surgery within the feet.The data was collected, grouped and analyzed separately for: PSSN, motor neuropathy (MN): MN-Calluses and MN-Feet deformity. One patient can developed PSSN and calluses and feet deformity (and thus his/her result was incorporated into each arm) or one of these variables.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Diabetes: Patients with diabetes from Diabetes Foot Center (DFC)
Arm/Group | Patients With Diabetes
Number analyzed (Participants) | 974
Participants
  PSSN: negative | 907
  PSSN: positive | 67
  MN calluses: negative | 645
  MN calluses: positive | 329
  MN feet deformity: negative | 798
  MN feet deformity: positive | 176

3. Secondary Outcome: BMI
Description: kg/m2
Time Frame: 1 visit
Population: Patients after BMI were assigned to one of two groups : BMI<35 kg/m2 or ≥35 kg/m2
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Diabetes: Patients with diabetes from DFC
Arm/Group | Patients With Diabetes
Number analyzed (Participants) | 974
Participants
  BMI ≥35 kg/m2 | 153
  BMI<35 kg/m2 | 821

ADVERSE EVENTS:
Time Frame: Not applicable- observational, retrospective study with medical-records analysis.
Description: Not applicable- observational, retrospective study with medical-records analysis.
Arm/Group | Patients With Diabetes
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Lack of the influence of a type and duration of diabetes mellitus.The neuropathy evaluation based on local recommendations.

The semi-quantitative analysis of the pressure map; the retrospective nature of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes